CLINICAL TRIAL: NCT02332824
Title: A Randomized, Multi-center, Double-blind, Placebo-controlled, Parallel-group Comparison, Phase 2 Study to Evaluate the Dose-response Relationship of the Efficacy and Safety of Oral Administration of TAK-272 in Patients With Type 2 Diabetes Mellitus and Microalbuminuria
Brief Title: A Phase 2 Dose-finding Study of TAK-272 in Participants With Type 2 Diabetes Mellitus and Microalbuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-272/CCT-101; JapicCTI-142658 (Registry Identifier: JapicCTI (Japan)); U1111-1161-6858 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2014-09-26; First posted 2015-01-07 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Mellitus and Microalbuminuria
Keywords: Pharmacological therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — imarikiren hydrochloride; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet orally, once daily for up to 12 weeks.
  Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
  Interventions: Drug: TAK-272 Placebo; Drug: Candesartan cilexetil Placebo
- TAK-272 5 mg (Experimental): TAK-272 5 mg one tablet, TAK-272 placebo 3 tablets and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks.
  Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
  Interventions: Drug: TAK-272; Drug: TAK-272 Placebo; Drug: Candesartan cilexetil Placebo
- TAK-272 20 mg (Experimental): TAK-272 20 mg one tablet, TAK-272 placebo 3 tablets and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks.
  Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
  Interventions: Drug: TAK-272; Drug: TAK-272 Placebo; Drug: Candesartan cilexetil Placebo
- TAK-272 40 mg (Experimental): TAK-272 20 mg 2 tablets, TAK-272 placebo 2 tablets, and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks.
  Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
  Interventions: Drug: TAK-272; Drug: TAK-272 Placebo; Drug: Candesartan cilexetil Placebo
- TAK-272 80 mg (Experimental): TAK-272 20 mg 4 tablets and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks.
  Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
  Interventions: Drug: TAK-272; Drug: Candesartan cilexetil Placebo
- Candesartan cilexetil 8 mg (Active Comparator): TAK-272 placebo 4 tablets and Candesartan cilexetil 8 mg one tablet, orally, once daily for up to 12 weeks.
  Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
  Interventions: Drug: TAK-272 Placebo; Drug: Candesartan cilexetil

INTERVENTIONS:
Drug: TAK-272 — TAK-272 tablets
  Arms: TAK-272 20 mg; TAK-272 40 mg; TAK-272 5 mg; TAK-272 80 mg
Drug: TAK-272 Placebo — TAK-272 placebo-matching tablets
  Arms: Candesartan cilexetil 8 mg; Placebo; TAK-272 20 mg; TAK-272 40 mg; TAK-272 5 mg
Drug: Candesartan cilexetil — Candesartan cilexetil tablets
  Arms: Candesartan cilexetil 8 mg
Drug: Candesartan cilexetil Placebo — Candesartan cilexetil placebo-matching tablets
  Arms: Placebo; TAK-272 20 mg; TAK-272 40 mg; TAK-272 5 mg; TAK-272 80 mg

SUMMARY:
The purpose of this study is to test the efficacy and safety on daily oral doses of TAK-272 5 mg, 20 mg, 40 mg and 80 mg in patients with type 2 diabetes mellitus and microalbuminuria by randomized, double-blind, placebo-controlled, parallel-group comparison in order to determine the clinical dose of TAK-272.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-272. This study evaluated the dose-response relationship of the efficacy and safety of TAK-272 in participants with type 2 diabetes mellitus and microalbuminuria.

The study enrolled 415 patients. Participants were randomly assigned to one of the 6 treatment groups:

* TAK-272 5 mg
* TAK-272 20 mg
* TAK-272 40 mg
* TAK-272 80 mg
* Candesartan cilexetil 8 mg
* Placebo (dummy inactive pill) for TAK-272 or Candesartan cilexetil - this was a tablet that looks like the study drug but had no active ingredient

All participants were administered tablets, orally at the same time each day for 12 weeks in double-blind manner. Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).

This multi-center trial was conducted in Japan. The overall time to participate in this study is 22 weeks including 2 weeks of follow-up assessment period after last dose of study drug. Participants made multiple visits to the clinic during these periods.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator or the sub-investigator, the participant is capable of understanding and complying with protocol requirements.
* The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
* The participant is either male or female and aged 20 to less than 75 years at signing of informed consent.
* The participant is an early-stage nephropathy (Stage 2) patient with type 2 diabetes mellitus.
* Inpatient/outpatient: outpatient
* The participant is a patient with type 2 diabetes mellitus on a certain diet therapy and/or exercise therapy (if any).
* The participant has stability controlled blood glucose, blood pressure and lipid, and does not need any change in the drug and the dose of any antihypertensive, antidiabetic and antidyslipidemia or antihyperlipidemic drugs throughout the study period as judged by the investigator or the sub-investigator.
* The participant has urine albumin/creatinine ratio (UACR) of the first morning urine (the first urine immediately after rising prior to activities in standing position in the morning) is ≥30 to <300 mg/gCr on at least two of three measurements at the start of the pre-treatment period (Week -8), at Week -4 or Week -2.
* The participant has estimated glomerular filtration rate according to creatinine (eGFRcreat) ≥45 mL/min/1.73 m^2 at Week -4.
* A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the study period and for 12 weeks after the completion of the study.
* A female participant of childbearing potential who is sexually active with a nonsterilized male partner who agrees to routinely use adequate contraception from signing of informed consent until 1 month after the completion of the study.

Exclusion Criteria:

<Exclusion Criteria in whole pre-treatment period>

* The participant received TAK-272 in a previous clinical study.
* The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent to participate under duress.
* The participant has a history of hypersensitivity or allergies to TAK-272, candesartan cilexetil and other renin-angiotensin system (RAS) inhibitors (angiotensin converting enzyme [ACE] inhibitors, angiotensin II receptor blocker [ARBs] or direct renin inhibitor [DRIs]).
* The participant needs to take the prohibited medications during the study period.
* The participant has hyperkalemia (e.g., serum potassium ≥ 5.0 mEq/L at the start of the pretreatment period (Week -8) and Week -4 or requiring regular use of a potassium adsorbent) or onset of hyperkalemia within 2 years prior to starting the pre-treatment period.
* The participant has at least class II hypertension (e.g., sitting systolic blood pressure [SBP] ≥160 mmHg or sitting diastolic blood pressure [DBP] ≥100 mmHg in the pre-treatment period) or malignant hypertension.
* The participant has a renal disease other than type 2 diabetic nephropathy (e.g., patients with renal sclerosis, acute or chronic glomerular nephritis, or polycystic kidney).
* The participant has bilateral or unilateral renal artery stenosis.
* The participant requires regular use of nonsteroidal anti-inflammatory drugs (excluding low-dose aspirin and locally-acting agents such as topical drugs) (e.g., rheumatoid arthritis patients, osteoarthritis patients, and low back pain patients).
* The participant has a history of any of the cardiovascular diseases listed below within 2 years prior to starting the pre-treatment period:

  * Cardiac diseases: myocardial infarction, coronary arterial revascularization
  * Cerebrovascular diseases: cerebral infarction (excluding lacunar infarction), cerebral hemorrhage, transient ischemic attack
* The participant has any of the cardiovascular diseases listed below:

  * Cardiac diseases: angina pectoris, arrhythmia, and congested heart failure that requires medication
  * Vascular diseases: arteriosclerosis obliterans with symptoms (e.g., intermittent claudication)
* The participant has a clinically significant hepatic disorder (e.g., either of alanine aminotransferase [ALT] or aspartate aminotransferase [AST] is ≥ 2.5 times the upper limit of normal at the start of the pre-treatment period (Week -8) or at Week -4).
* The participant has a complication of malignant tumor.
* If female, the participant is pregnant, lactating, or is intending to become pregnant before, during or within 1 month after participating in this study; or intending to donate ova during such time period.
* If male, the participant intends to donate sperm during the course of this study or for 12 weeks thereafter.
* The participant is judged by the investigator or the sub-investigator as being ineligible for any other reason.

<Exclusion Criteria at the start of the pre-treatment period (Week -8)>

* The participant has participated in another clinical study or post-marketing study within 30 days prior to starting the pre-treatment period.
* The participant has received the study medication within 12 weeks prior to starting the pre-treatment period.
* The participant has a history of drug abuse (defined as the use of an illicit drug) or history of alcohol abuse within 2 years prior to starting the pre-treatment period.
* The participant has changed the renin angiotensin system (RAS) inhibitor (angiotensin-converting enzyme [ACE] inhibitor, angiotensin II receptor blocker [ARB] or direct renin inhibitors [DRI]) or its dose and regimen within 12 weeks prior to starting the pre-treatment period.
* The participant is treated with any RAS inhibitor (ACE inhibitor, ARB or DRI) at signing of informed consent, and whose UACR is <30 mg/gCr at the start of the pre-treatment period (Week -8).

<Exclusion Criteria at Week -4>

* The participant has hemoglobin A1c (HbA1c) (National Glycohemoglobin Standardization Program [NGSP]) ≥9.0% at Week -4.
* The participant has change in HbA1c (NGSP) from the start of the pre-treatment period (Week -8) to Week -4 by ≥10.0%* compared to the higher value of them.

  *Second decimal place to be rounded off <Exclusion Criteria at the end of the Pre-treatment period (Week 0)>
* The participant's sitting SBP and sitting DBP changed by ≥20 mmHg or ≥10 mmHg, respectively, at the end of the pre-treatment period (Week 0) compared to Week -2.
* The participant's sitting SBP is <130 mmHg at the end of the pre-treatment period (Week 0).
* The participant's study drug compliance rate* during the pre-treatment period is <80.0%.

  * Compliance rate (%)=(Prescribed amount-Retrieved amount)/ {(Completion date of study drug for the pre-treatment period-Starting date of study drug for the pre-treatment period+1)×5}×100, second decimal place to be rounded off.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (68):
- Japan (68):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Kisarazu-shi, Chiba
  - Fukuoka, Fukuoka
  - Fukutsu-shi, Fukuoka
  - Kitakyuushu-shi, Fukuoka
  - Kouriyama-shi, Fukushima
  - Anchu-shi, Gunma
  - Ota-shi, Gunma
  - Ishikari-shi, Hokkaido
  - Obihiro-shi, Hokkaido
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Moriya-shi, Ibaragi
  - Naka, Ibaragi
  - Koga, Ibarakgi
  - Koga-shi, Ibaraki
  - Mito, Ibaraki
  - Takamatsu, Kagawa-ken
  - Ebina-shi, Kanagawa
  - Hiratsuka-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Miura-shi, Kanagawa
  - Shounann-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Yatsushiro-shi, Kumamoto
  - Kyoto, Kyoto
  - Uji-shi, Kyoto
  - Sendai, Miyagi
  - Miyazaki, Miyazaki
  - Azumino-shi, Nagano
  - Matsumoto-shi, Nagano
  - Nakano-shi, Nagano
  - Sasebo-shi, Nagasaki
  - Kasaoka-shi, Okayama-ken
  - Kurashiki-shi, Okayama-ken
  - Naha, Okinawa
  - Shimajiri-gun, Okinawa
  - Tomigusuku-shi, Okinawa
  - Kashiwara-shi, Osaka
  - Matsubara-shi, Osaka
  - Neyagawa, Osaka
  - Osaka, Osaka
  - Suita-shi, Osaka
  - Tondabayashi-shi, Osaka
  - Kawagoe-shi, Saitama
  - Kyuki-shi, Saitama
  - Saitama-shi, Saitama
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Koyama-shi, Tochigi
  - Shimono-shi, Tochigi
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Hachioji-shi, Tokyo
  - Hino-shi, Tokyo
  - Itabashi-ku, Tokyo
  - Katsushika-ku, Tokyo
  - Nerima-ku, Tokyo
  - Ōta-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Shinjyuku-ku, Tokyo
  - Ube-shi, Yamaguchi

REFERENCES:
- [Derived] Wang GM, Li LJ, Fan L, Xu M, Tang WL, Wright JM. Renin inhibitors versus angiotensin receptor blockers for primary hypertension. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD012570. doi: 10.1002/14651858.CD012570.pub2. PMID 40013543

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 81 investigative sites in Japan from 16 Oct 2014 to 18 Aug 2016.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes mellitus and microalbuminuria (early-stage nephropathy [Stage 2] patients with type 2 diabetes mellitus) were randomized in 1:1:1:1:1:1 to either of TAK-272 5 mg, 20 mg, 40 mg, 80 mg, candesartan cilexetil 8 mg or Placebo and administered tablets orally once daily for 12 weeks in double-blind manner.
Groups:
- Placebo: TAK-272 placebo, 4 tablets, and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks. Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
- TAK-272 5 mg: TAK-272 5 mg, one tablet, TAK-272 placebo 3 tablets, and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks. Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
- TAK-272 20 mg: TAK-272 20 mg, one tablet, TAK-272 placebo 3 tablets, and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks. Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
- TAK-272 40 mg: TAK-272 20 mg, 2 tablets, TAK-272 placebo 2 tablets, and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks. Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
- TAK-272 80 mg: TAK-272 20 mg, 4 tablets, and Candesartan cilexetil placebo one tablet, orally, once daily for up to 12 weeks. Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
- Candesartan Cilexetil 8 mg: Candesartan cilexetil 8 mg, one tablet, and TAK-272 placebo 4 tablets, orally, once daily for up to 12 weeks. Participants were administered TAK-272 placebo 4 tablets and Candesartan cilexetil placebo one tablet for 4 weeks (Week -4 to 0) in placebo run-in period and follow-up period (Week 12-14).
Period: Overall Study
Arm/Group | Placebo | TAK-272 5 mg | TAK-272 20 mg | TAK-272 40 mg | TAK-272 80 mg | Candesartan Cilexetil 8 mg
Started | 67 | 67 | 74 | 68 | 69 | 70
Completed | 61 | 66 | 72 | 66 | 65 | 69
Not Completed | 6 | 1 | 2 | 2 | 4 | 1
Not completed — Pretreatment Event/Adverse Event | 4 | 0 | 1 | 1 | 4 | 1
Not completed — Voluntary Withdrawal | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Inconvenient schedule | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Transfer | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-272 5 mg | TAK-272 20 mg | TAK-272 40 mg | TAK-272 80 mg | Candesartan Cilexetil 8 mg | Total
Number analyzed (Participants) | 67 | 67 | 74 | 68 | 69 | 70 | 415
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.38) | 61.8 (8.90) | 60.9 (9.57) | 59.6 (10.22) | 61.2 (9.95) | 62.4 (9.29) | 61.3 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 17 | 13 | 18 | 14 | 89
  Male | 51 | 56 | 57 | 55 | 51 | 56 | 326
Region of Enrollment [Number; unit: participants] — All participants were enrolled in Japan.
  participants
    Japan | 67 | 67 | 74 | 68 | 69 | 70 | 415
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]. Population: The analyzed numbers for each arm were participants who were evaluable for this baseline characteristic.
  kg/m^2
    number analyzed (Participants) | 67 | 67 | 73 | 68 | 69 | 70 | 414
    (all) | 25.93 (4.024) | 26.41 (4.208) | 26.91 (5.035) | 26.39 (4.580) | 26.41 (3.543) | 26.60 (5.483) | 26.45 (4.518)
Duration of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: years] | 12.24 (8.164) | 11.48 (7.355) | 11.06 (7.708) | 11.19 (7.151) | 10.88 (7.363) | 10.38 (7.046) | 11.19 (7.450)
Concurrent Medical Condition [Count of Participants; unit: Participants] — Participants may also be counted in more than 1 category.
  Participants
    Hypertension - Yes | 50 | 46 | 60 | 48 | 60 | 52 | 316
    Hypertension - No | 17 | 21 | 14 | 20 | 9 | 18 | 99
    Dyslipidemia - Yes | 45 | 41 | 58 | 51 | 56 | 46 | 297
    Dyslipidemia - No | 22 | 26 | 16 | 17 | 13 | 24 | 118
Previous Medication [Count of Participants; unit: Participants] — Participants may also be counted in more than 1 category.
  Participants
    Renin-angiotensin system (RAS) Inhibitor - Yes | 30 | 31 | 33 | 25 | 36 | 35 | 190
    RAS Inhibitor - No | 37 | 36 | 41 | 43 | 33 | 35 | 225
    Sodium Glucose Co-transporter (SGLT2)Inhibitor-Yes | 1 | 2 | 3 | 1 | 2 | 0 | 9
    SGLT2 Inhibitor - No | 66 | 65 | 71 | 67 | 67 | 70 | 406
    Potassium-Sparing Diuretic - Yes | 0 | 1 | 0 | 1 | 0 | 1 | 3
    Potassium-Sparing Diuretic - No | 67 | 66 | 74 | 67 | 69 | 69 | 412
Restricted Medication [Count of Participants; unit: Participants] — HMG-COA = 3-hydroxy-3-methylglutaryl Coenzyme A. Participants may also be counted in more than 1 category.
  Participants
    Anti-Hypertension Drug - Yes | 40 | 34 | 46 | 33 | 44 | 45 | 242
    Anti-Hypertension Drug - No | 27 | 33 | 28 | 35 | 25 | 25 | 173
    Anti-Diabetic Drug - Yes | 64 | 64 | 66 | 65 | 65 | 66 | 390
    Anti-Diabetic Drug - No | 3 | 3 | 8 | 3 | 4 | 4 | 25
    HMG-CoA Reductase Inhibitor - Yes | 30 | 27 | 35 | 31 | 44 | 27 | 194
    HMG-CoA Reductase Inhibitor - No | 37 | 40 | 39 | 37 | 25 | 43 | 221
Urine albumin/Creatinine ratio [Median (Inter-Quartile Range); unit: mg/gCR] — Population: The analyzed numbers for each arm were participants who were evaluable for this baseline characteristic.
  mg/gCR
    number analyzed (Participants) | 67 | 67 | 73 | 68 | 69 | 70 | 414
    (all) | 119.95 [65.61 to 214.88] | 93.45 [53.92 to 139.41] | 96.03 [58.59 to 174.45] | 116.43 [49.92 to 201.16] | 86.87 [53.53 to 153.05] | 96.33 [57.48 to 179.26] | 100.26 [55.90 to 179.37]
eGFRcreat [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Male: eGFRcreat (mL/min/1.73 m^2)=194×Cr (mg/dL)^(-1.094)×age (years)^(-0.287) Female: eGFRcreat (mL/min/1.73 m^2)=194×Cr (mg/dL)^(-1.094)×age (years)^(-0.287)×0.739 Cr: serum creatinine Population: The analyzed numbers for each arm were participants who were evaluable for this baseline characteristic.
  mL/min/1.73m^2
    number analyzed (Participants) | 67 | 67 | 72 | 68 | 69 | 70 | 413
    (all) | 77.17 (18.828) | 81.81 (19.788) | 79.19 (19.449) | 80.51 (20.292) | 77.81 (18.425) | 83.27 (22.777) | 79.97 (19.980)
Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycated haemoglobin] — Population: The analyzed numbers for each arm were participants who were evaluable for this baseline characteristic.
  percentage of glycated haemoglobin
    number analyzed (Participants) | 67 | 67 | 73 | 68 | 69 | 70 | 414
    (all) | 7.02 (0.789) | 7.03 (0.772) | 7.06 (0.770) | 7.03 (0.789) | 6.90 (0.834) | 7.02 (0.731) | 7.01 (0.778)
Trough Sitting Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: The analyzed numbers for each arm were participants who were evaluable for this baseline characteristic.
  mmHg
    number analyzed (Participants) | 67 | 67 | 73 | 68 | 69 | 70 | 414
    (all) | 80.6 (9.29) | 80.6 (8.80) | 80.6 (8.99) | 79.3 (9.26) | 81.9 (8.90) | 80.5 (8.89) | 80.6 (9.00)
Trough Sitting Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: The analyzed numbers for each arm were participants who were evaluable for this baseline characteristic.
  mmHg
    number analyzed (Participants) | 67 | 67 | 73 | 68 | 69 | 70 | 414
    (all) | 141.1 (7.01) | 139.0 (8.41) | 138.2 (7.09) | 139.0 (7.64) | 140.3 (7.77) | 140.6 (7.65) | 139.7 (7.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From End of Pre-treatment Period (Week 0) in Log-transformed Urine Albumin/Creatinine Ratio (UACR) at the End of Treatment Period (Week 12)
Description: The first morning void urine (the first urine immediately after rising prior to activities in standing position in the morning) samples on the day of each visit, and 1 day and 2 days before the day of each visit (3 consecutive days) were collected to calculate UACR.
Time Frame: Week 0 and Week 12
Population: Full analysis set (FAS) included all participants who were randomized and received at least one dose of the study drug for the treatment period. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: log (mg/gCr)
Arm/Group | Placebo | TAK-272 5 mg | TAK-272 20 mg | TAK-272 40 mg | TAK-272 80 mg | Candesartan Cilexetil 8 mg
Number analyzed (Participants) | 66 | 67 | 73 | 67 | 69 | 70
log (mg/gCr) | 0.152 [0.0389 to 0.2655] | -0.173 [-0.2848 to -0.0602] | -0.317 [-0.4245 to -0.2095] | -0.478 [-0.5904 to -0.3661] | -0.497 [-0.6081 to -0.3867] | -0.377 [-0.4872 to -0.2678]
Statistical Analysis 1: Comparison: Placebo vs TAK-272 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — In the primary analysis, each TAK-272 group will be compared with placebo group based on a step-down testing procedure, which will be employed for multiple comparison adjustment; LS Mean difference = -0.325, 95% CI 2-sided [-0.4845 to -0.1649] — Estimated Value was for LS mean differences (TAK-272 5 mg-placebo) in log-transformed UACR changes from baseline to the end of treatment period
Statistical Analysis 2: Comparison: Placebo vs TAK-272 20 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean difference = -0.469, 95% CI 2-sided [-0.6251 to -0.3132] — Estimated Value was for LS mean differences (TAK-272 20 mg-placebo) in log-transformed UACR changes from baseline to the end of treatment period
Statistical Analysis 3: Comparison: Placebo vs TAK-272 40 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean difference = -0.630, 95% CI 2-sided [-0.7897 to -0.4711] — Estimated Value was for LS mean differences (TAK-272 40 mg -placebo) in log-transformed UACR changes from baseline to the end of treatment period
Statistical Analysis 4: Comparison: Placebo vs TAK-272 80 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean difference = -0.650, 95% CI 2-sided [-0.8083 to -0.4908] — Estimated Value was for LS mean differences (TAK-272 80 mg -placebo) in log-transformed UACR changes from baseline to the end of treatment period
Statistical Analysis 5: Comparison: Placebo vs Candesartan Cilexetil 8 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean difference = -0.530, 95% CI 2-sided [-0.6874 to -0.3719] — Estimated Value was for LS mean differences (Candesartan cilexetil 8 mg -placebo group) in log-transformed UACR changes from baseline to the end of treatment period

2. Secondary Outcome: Urine Albumin/Creatinine Ratio (UACR) at Each Assessment Point
Description: The first morning void urine (the first urine immediately after rising prior to activities in standing position in the morning) samples on the day of each visit, and 1 day and 2 days before the day of each visit (3 consecutive days) were collected to calculate UACR. Reported data is geometric mean ratio of UACR at each assessment point relative to Baseline.
Time Frame: Weeks 2, 4, 8, 12, follow-up (Week 14) and End of Treatment
Population: The FAS included all participants who were randomized and received at least one dose of the study drug for the treatment period. The analyzed numbers for each arm were participants who were evaluable for this outcome measure at particular timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/gCr
Arm/Group | Placebo | TAK-272 5 mg | TAK-272 20 mg | TAK-272 40 mg | TAK-272 80 mg | Candesartan Cilexetil 8 mg
Number analyzed (Participants) | 67 | 67 | 74 | 68 | 69 | 70
mg/gCr
  Week 2: number analyzed (Participants) | 66 | 67 | 73 | 66 | 69 | 70
  Week 2 | 1.04 [0.979 to 1.112] | 0.84 [0.767 to 0.929] | 0.80 [0.736 to 0.873] | 0.73 [0.678 to 0.795] | 0.72 [0.659 to 0.797] | 0.76 [0.708 to 0.812]
  Week 4: number analyzed (Participants) | 65 | 67 | 73 | 67 | 68 | 70
  Week 4 | 1.03 [0.930 to 1.132] | 0.82 [0.742 to 0.901] | 0.80 [0.731 to 0.881] | 0.66 [0.605 to 0.722] | 0.71 [0.638 to 0.781] | 0.72 [0.668 to 0.782]
  Week 8: number analyzed (Participants) | 64 | 67 | 71 | 66 | 65 | 70
  Week 8 | 1.07 [0.974 to 1.182] | 0.85 [0.772 to 0.942] | 0.75 [0.686 to 0.817] | 0.63 [0.569 to 0.688] | 0.62 [0.552 to 0.690] | 0.71 [0.639 to 0.786]
  Week 12: number analyzed (Participants) | 61 | 67 | 71 | 66 | 65 | 69
  Week 12 | 1.13 [1.025 to 1.238] | 0.85 [0.760 to 0.947] | 0.71 [0.631 to 0.793] | 0.61 [0.546 to 0.685] | 0.59 [0.519 to 0.672] | 0.70 [0.630 to 0.776]
  Follow-up (Week 14): number analyzed (Participants) | 60 | 65 | 71 | 65 | 63 | 69
  Follow-up (Week 14) | 1.11 [0.985 to 1.255] | 0.92 [0.830 to 1.031] | 0.95 [0.861 to 1.055] | 0.80 [0.725 to 0.872] | 0.86 [0.770 to 0.966] | 0.85 [0.771 to 0.936]
  End of treatment: number analyzed (Participants) | 66 | 67 | 73 | 67 | 69 | 70
  End of treatment | 1.15 [1.048 to 1.267] | 0.85 [0.760 to 0.947] | 0.72 [0.644 to 0.815] | 0.62 [0.552 to 0.693] | 0.61 [0.540 to 0.698] | 0.69 [0.616 to 0.765]

3. Secondary Outcome: Remission Rate From Early-Stage Nephropathy (Stage 2) to Pre-Nephropathy Stage (Stage 1) at the End of Treatment (Week 12)
Description: Remission rate is defined as percentage of participants who have UACR <30 mg/gCr and whose UACR decreased by ≥30% from the value at the end of the pre-treatment period (Week 0).
Time Frame: Week 12
Population: The FAS included all participants who were randomized and received at least one dose of the study drug for the treatment period. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-272 5 mg | TAK-272 20 mg | TAK-272 40 mg | TAK-272 80 mg | Candesartan Cilexetil 8 mg
Number analyzed (Participants) | 66 | 67 | 74 | 67 | 69 | 70
percentage of participants | 0.0 [0.000 to 5.436] | 9.0 [3.358 to 18.480] | 9.5 [3.888 to 18.524] | 17.9 [9.612 to 29.196] | 24.6 [15.055 to 36.490] | 14.3 [7.069 to 24.707]

4. Secondary Outcome: Progression Rate From Early-Stage Nephropathy (Stage 2) to Overt Nephropathy (Stage 3) During the Treatment Period (Week 12)
Description: Progression rate is defined as percentage of participants who have UACR ≥300 mg/gCr and whose UACR increased by ≥30% from the value at the end of the pre-treatment period [Week 0]. Meanwhile, the definition of transition to overt nephropathy also includes the case that UACR decreased to <300 mg/gCr after the transition to overt nephropathy.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-272 5 mg | TAK-272 20 mg | TAK-272 40 mg | TAK-272 80 mg | Candesartan Cilexetil 8 mg
Number analyzed (Participants) | 66 | 67 | 74 | 67 | 69 | 70
percentage of participants | 18.2 [9.764 to 29.607] | 3.0 [0.364 to 10.371] | 0.0 [0.000 to 4.863] | 0.0 [0.000 to 5.357] | 0.0 [0.000 to 5.206] | 1.4 [0.036 to 7.704]

5. Other Pre Specified Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to Week 14
Population: Safety analysis set included all participants who received at least one dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-272 5 mg | TAK-272 20 mg | TAK-272 40 mg | TAK-272 80 mg | Candesartan Cilexetil 8 mg
Number analyzed (Participants) | 67 | 67 | 74 | 68 | 69 | 70
Participants | 28 | 22 | 26 | 28 | 36 | 30

ADVERSE EVENTS:
Time Frame: Up to Week 14
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-272 5 mg | TAK-272 20 mg | TAK-272 40 mg | TAK-272 80 mg | Candesartan Cilexetil 8 mg
Serious Adverse Events (participants affected / at risk) | 2/67 | 0/67 | 0/74 | 0/68 | 2/69 | 1/70
Other Adverse Events (participants affected / at risk) | 7/67 | 7/67 | 8/74 | 9/68 | 11/69 | 11/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | TAK-272 5 mg (N=67) | TAK-272 20 mg (N=74) | TAK-272 40 mg (N=68) | TAK-272 80 mg (N=69) | Candesartan Cilexetil 8 mg (N=70)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | TAK-272 5 mg (N=67) | TAK-272 20 mg (N=74) | TAK-272 40 mg (N=68) | TAK-272 80 mg (N=69) | Candesartan Cilexetil 8 mg (N=70)
Nasopharyngitis (Infections and infestations) | 7 | 7 | 8 | 9 | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.